CLINICAL TRIAL: NCT01262664
Title: A First-in-Man, Phase I Evaluation of A Single Cycle of Prohibitin Targeting Peptide 1 in Patients With Metastatic Prostate Cancer and Obesity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0369; NCI-2011-00300 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Advanced prostate cancer; Castrate-Resistant Prostate Cancer; Prohibitin-TP01
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prohibitin-TP01 (Experimental): Prohibitin-TP01 starting dose of 0.03 mg/kg as an injection under the skin 1 time each day for 28 days.
  Interventions: Drug: Prohibitin-TP01

INTERVENTIONS:
Drug: Prohibitin-TP01 — Starting dose of 0.03 mg/kg as an injection under the skin 1 time each day for 28 days.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of PROHIBITIN-TP01 that can be given to patients with advanced prostate cancer for which there are no standard therapy options. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

PROHIBITIN-TP01 is designed to destroy "white fat" (the type of fat that collects around the stomach and is associated with obesity in men). Fat is known to produce substances that can promote prostate cancer growth. Investigators want to learn if decreasing fat can slow the growth of prostate cancer.

This is the first study using PROHIBITIN-TP01 in humans.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of PROHIBITIN-TP01 based on when you join this study. Up to 5 dose levels of PROHIBITIN-TP01 will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of PROHIBITIN-TP01 is found.

Study Drug Administration:

You will receive PROHIBITIN-TP01 as an injection under the skin 1 time each day for 28 days.

Study Visits:

On Days 1, 8, 15 and 22:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests. You will be required to fast for about 8 hours before this blood test.
* You will be asked about any symptoms or side effects you may have had since your last visit and about any other drugs you may be taking.
* Blood (about 2 teaspoons) will be drawn for PK testing 10 minutes, 30 minutes, 1 hour, and 4 hours after you receive the Day 1 and Day 22 dose of PROHIBITIN-TP01.
* You will have an ECG either right before or within 4 hours after you receive the study drug (Days 1, 15, and 22 only).

Length of Study Drug Administration:

You will receive the study drug for up to 28 days. You will no longer be able to receive the study drug if the disease gets worse or intolerable side effects occur.

Follow-up Visit:

Within 7 days after you stop receiving the study drug, the following procedures will be performed:

* You will have a physical exam, including measurement of your weight, as well as measurements of your waist and hips.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests. This testing will also include a measurement of your PSA, testosterone, cholesterol, and other research tests that may show how the study drug affected you.
* You will be asked about symptoms or any side effects you have had since your last visit.
* You will have CT or MRI scans and a chest x-ray to check the status of the disease.
* You will have an ECG

Thirty (30) days after you stop receiving the study drug, the following procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* Blood (about 3 teaspoons - in addition to that listed above) will be collected to learn if your immune system reacts to PROHIBITIN-TP01 by forming antibodies.
* You will be asked about symptoms or any side effects you have had since your last visit.
* You will have an ECG

Long-Term Follow-Up:

You will be contacted by phone or e-mail every 3 months for 1 year and asked about your kidney function, current weight, prostate cancer status, and any side effects you may have had. Each phone call will last up to 5 minutes.

This is an investigational study. PROHIBITIN-TP01 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 39 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed carcinoma of the prostate that is metastatic or otherwise incurable, and a BMI defined as obese (i.e. >30 kg/m2). Any histologic variant is acceptable other than small cell carcinoma.
2. Have been on androgen deprivation therapy for a minimum of 6 months, and continue that therapy or an equivalent therapy to suppress testosterone during this trial.
3. Patients with castrate resistant prostate cancer (CRPC) must have no standard options for therapy. Prior to registration on the study, patients with CRPC must be at least 3 weeks from their last treatment, such as ketoconazole, abiraterone, low-dose dexamethasone, anti-androgens, or cytotoxic therapy, (excluding ongoing therapy to suppress testosterone, which must also be continued during this trial).
4. Have an ECOG performance status 0, 1 or 2
5. Have adequate bone marrow function defined as an absolute peripheral granulocyte count of >/= 1,000/mm^3 and platelet count of >/= 100,000/mm^3; hemoglobin >/= 8.0 g/dL (without transfusion or growth factor support)
6. Have adequate hepatic function defined as a total bilirubin of </= 1.5 mg/dl and AST </= 2x the upper limits of normal
7. Have adequate renal function defined as serum creatinine </= 1.5x the upper limit of normal or creatinine clearance >/= 60 mL/min (measured or calculated). In addition, patients must have a 24 hr urine collection showing less than 2000 mg of protein. EXCEPTION: Patients with hematuria will be eligible with up to 3000 mg protein per 24 hours provided they do not have casts, eosinophiluria or electrolyte wasting.
8. Have adequate cardiovascular function as defined by: i) a normal B-type Natruetic Peptide (BNP) with ii) no signs or symptoms suggestive of cardiac disease and iii) a normal ECG. If these criteria are not met, patients must have an echocardiogram or multigated cardiac scan (MUGA) showing an EF of 45% or greater with no more than "mild" diastolic dysfunction and a BNP of < 200 pg/mL to be eligible.
9. Sign the current IRB approved informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution

Exclusion Criteria:

1. Small cell prostate cancer
2. Infectious process, which, in the opinion of the investigator, could worsen or its outcome be affected, as a result of the investigational therapy
3. Any of the following in previous 6 months: NYHA Class III/IV congestive heart failure, unstable angina, cerebrovascular accident (including transient ischemic attack), pulmonary embolism or myocardial infarction (by ECG or serologic criteria)
4. Significant co-morbidity that could affect the safety or evaluability of participants, specifically including: i) Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 140 or diastolic pressures above 90 despite therapy. Note that this may be better established with home BP readings than with clinic visit results. Note further that this is NOT a criterion related to particular BP results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes. The intent is to exclude patients that may have unrecognized renal damage from chronic, uncontrolled hypertension, NOT to exclude patients who may be hypertensive acutely. There are no absolute criteria for BP readings with respect to eligibility (as determined by treating physician).
5. ( # 9 cont'd) (ii) Uncontrolled diabetes mellitus, defined as: Hgb A1c >8.5%; or symptomatic hypoglycemic episodes > 1 per week during the two months prior to eligibility evaluation; or more than 1 glucose excursion to >300 mg/dL in prior two months--unless clearly iatrogenic and the cause has been eliminated iii) Lung disease requiring supplemental oxygen iv) Known chronic liver disease causing either fibrosis or synthetic dysfunction v) Known HIV infection vi) Overt psychosis, mental disability or being otherwise incompetent to grant informed consent or a history of non-compliance with medical care.
6. Hydronephrosis (either bilateral or involving a solitary kidney) that has not been addressed by means of a nephrostomy or indwelling stent. EXCEPTION: Non-obstructive hydronephrosis in setting of prior urinary diversion is consistent with eligibility.
7. Patients require ongoing therapy with non-steroidal anti-inflammatory drugs (NSAIDs), i.v. vancomycin, aminoglycosides, or other potently nephrotoxic drugs, and must agree to abstain from NSAIDs from the time the consent is signed up until 30 days after the last dose of study drug is received, other than low-dose aspirin (81 mg/day or less).
8. Any other medical condition that in the opinion of the principal investigator would compromise the ability to deliver or evaluate study drug.
9. Unwillingness to maintain adequate contraception measures for the entire course of the study
10. Age < 18 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-05-24 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Acceptable Dose of Prohibitin-TP01 in Participants with Metastatic Prostate Cancer and Obesity | 58 days
  Dose is acceptable if is not unlikely that a dose has at least a 50% response rate, and that it is not unlikely that the dose has at most a 30% toxicity rate.
Biologic Activity of Prohibitin-TP01 in Participants with Metastatic Prostate Cancer and Obesity | 28 days
  Biologic Activity (BA) defined as loss of 10% of baseline body weight (or equivalently, a 10% reduction in BMI) as measured at the end of the 28 day dosing period.

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org